CLINICAL TRIAL: NCT06356714
Title: An Open Intervention Study of Nocardia Rubra Cell Wall Skeleton in Combination With Prior Second- or Third-line Regimens for the Treatment of Potentially Hazardous Colorectal Cancer SD(Stable Disease) Status
Brief Title: Nocardia Rubra Cell Wall Skeleton in Combination With Prior Second- or Third-line Regimens for the Treatment of Potentially Hazardous Colorectal Cancer SD Status
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Jing (Other)
Responsible Party: Sponsor-Investigator, Sun Jing, chief physician、professor, The First Affiliated Hospital with Nanjing Medical University
Organization: The First Affiliated Hospital with Nanjing Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13914704179
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms
Keywords: Nocardia Rubra Cell Wall Skeleton; Colorectal Cancer; Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nocardia Rubra Cell Wall Skeleton +prior Second- or Third-line Regimens (Experimental): The patient has previously received second- or third-line treatment for advanced or metastatic colorectal cancer and has developed a potentially hazardous SD (Stable Disease) status. They will add to the original treatment regimen of Nocardia Rubra Cell Wall Skeleton.
  Interventions: Drug: Nocardia Rubra Cell Wall Skeleton in Combination With Prior Second- or Third-line Regimens

INTERVENTIONS:
Drug: Nocardia Rubra Cell Wall Skeleton in Combination With Prior Second- or Third-line Regimens — Nocardia Rubra Cell Wall Skeleton 200 mcg-400 mcg, 0.3 ml diluted in water for injection or lidocaine, was injected subcutaneously every 2 or 3 weeks.
  Efficacy was evaluated every 2 cycles according to RECIST 1.1 criteria. Patients are enrolled and given this study regimen of drugs on top of their prior second- or third-line regimen until disease progression or intolerable toxicities occur; or the patient requests to be discharged.

SUMMARY:
Evaluate the efficacy and safety of Nocardia rubra cell wall skeleton in combination with prior second- or third-line regimens for the treatment of potentially hazardous colorectal cancer SD(Stable Disease) status in the real world.

DETAILED DESCRIPTION:
This is a prospective interventional clinical trial investigating the efficacy and safety of Nocardia rubra cell wall skeleton in combination with prior second- or third-line regimens for the treatment of potentially hazardous colorectal cancer SD (Stable Disease) status in the real world.

Enrollment requirements were patients who had received prior second- or third-line therapy for advanced or metastatic colorectal cancer and presented with a potentially harmful SD status.

The potentially hazardous SD (Stable Disease) state is defined as an increase in SLD (Sum of Longest Diameters) by less than 20% according to RECIST 1.1 criteria, with an absolute increase of SLD ≤ 5mm from the nadir; a serum CEA (Carcinoembryonic Antigen) level below 10.0 ng/ml during stable disease, with two consecutive measurements of 10 ng/ml or more (with a testing interval of at least one month); or a serum CEA level of 10 ng/ml or more during stable disease, with a gradual increase in CEA after two consecutive measurements (with a testing interval of at least one month); a serum CA19-9 level below 60.0 ng/ml during stable disease, with two consecutive measurements of 60 ng/ml or more (with a testing interval of at least one month); or a serum CEA level of 60 ng/ml or more during stable disease, with a gradual increase in CEA after two consecutive measurements (with a testing interval of at least one month). Meeting any one of the above criteria can be considered as the presence of a potentially hazardous SD state.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, gender is not limited;
2. Colorectal adenocarcinoma confirmed by pathologic histology and/or cytology and imaging;
3. Have 1 or more measurable lesions with a longest diameter of at least 10 mm as determined by spiral CT scanning; and a diameter of at least 20 mm as determined by conventional CT scanning (Criteria for the Evaluation of Efficacy in Solid Tumors, i.e., RECIST Criteria, version 1.1);
4. Prior second- or third-line therapy for advanced or metastatic colorectal cancer with potentially harmful SD status. The potentially hazardous SD (Stable Disease) state is defined as an increase in SLD (Sum of Longest Diameters) by less than 20% according to RECIST 1.1 criteria, with an absolute increase of SLD ≤ 5mm from the nadir; a serum CEA (Carcinoembryonic Antigen) level below 10.0 ng/ml during stable disease, with two consecutive measurements of 10 ng/ml or more (with a testing interval of at least one month); or a serum CEA level of 10 ng/ml or more during stable disease, with a gradual increase in CEA after two consecutive measurements (with a testing interval of at least one month); a serum CA19-9 level below 60.0 ng/ml during stable disease, with two consecutive measurements of 60 ng/ml or more (with a testing interval of at least one month); or a serum CEA level of 60 ng/ml or more during stable disease, with a gradual increase in CEA after two consecutive measurements (with a testing interval of at least one month). Meeting any one of the above criteria can be considered as the presence of a potentially hazardous SD state.
5. The general condition score of the Eastern Cooperative Oncology Group (ECOG) is 0 or 1;
6. Expected survival ≧3 months;
7. Blood, liver and kidney function within 7 days prior to screening: absolute neutrophil count ≥ 1.5 x 109 /L; hemoglobin ≥ 9.0 g/dl; platelet count ≥ 100 x 109 /L; total bilirubin ≤ 1.5 times the upper limit of normal (ULN); gammaglutaminase and gammaglutaminase ≤ 3.0 x ULN (≤ 5 x ULN for patients with hepatic metastases); alkaline phosphatase ≤ 3 x ULN. phosphatase ≤ 3 x ULN (≤ 5 x ULN in patients with liver metastases); serum creatinine ≤ 1.5 x ULN;
8. Agreed to sign the informed consent form;

Exclusion Criteria:

1. Allergic constitution;
2. With comorbid diabetes;
3. Active clinically severe infection;
4. Any other conditions deemed exclusionary by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2026-09-24 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | 1 year
  Time between the start of a treatment regimen and tumor progression or death

SECONDARY OUTCOMES:
Overall survival (OS) | 2 year
Objective remission rate (ORR) | 1 year
Disease Control Rate (DCR) | 1 year
Incidence and extent of major security incidents | 1 year
Quality of Life Score (QoL) for tumor patients | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No